CLINICAL TRIAL: NCT05398848
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled Phase III Trial to Evaluate the Efficacy, Safety and Immunogenicity of the Recombinant Two-component COVID-19 Vaccine (CHO Cell) in Adults Aged 18 Years and Older
Brief Title: Efficacy, Safety and Immunogenicity Study of the Recombinant Two-component COVID-19 Vaccine (CHO Cell)(Recov)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Rec-Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REC611C303
Record Dates: First submitted 2022-05-30; First posted 2022-06-01 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant two-component COVID-19 vaccine (CHO cell) (Experimental): Antigen: NTD-RBD-foldon protein, Adjuvant (BFA03)
  Interventions: Biological: Recombinant two-component COVID-19 vaccine (CHO cell)
- Placebo (Placebo Comparator): Adjuvant (BFA03)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant two-component COVID-19 vaccine (CHO cell) — Before reconstitution: Lyophilized powder for reconstitution in single-use vials After reconstitution with BFA03 adjuvant: Milk-white solution with no visible foreign matter
  Arms: Recombinant two-component COVID-19 vaccine (CHO cell)
Biological: Placebo — Before reconstitution:
  Lyophilized powder for reconstitution in single-use vials
  After reconstitution with BFA03 adjuvant:
  Milk-white solution with no visible foreign matter
  Arms: Placebo

SUMMARY:
This is a multicenter designed Phase III clinical trial. About 10000 participants plan to be enrolled.The objectives of this study are to evaluate the efficacy, safety and immunogenicity of the recombinant two-component COVID-19 vaccine (CHO cell) in adults

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blinded, placebo-controlled Phase III clinical trial. The objectives are to evaluate the efficacy, safety, and immunogenicity of ReCOV in adults aged 18 years and older who have not received any COVID-19 vaccination, and have no history of known COVID-19 in previous 6 months. Three-dose intramuscular (IM) vaccination schedule (21 days interval) will be applied.

About 10000 participants (about 15% participants ≥ 60 years old) with SARS-CoV-2 antibody (IgM and IgG) negative at baseline, will be randomized in a ratio of 1:1 to receive ReCOV (20 μg) or placebo on Day 0, Day 21, and Day 42, respectively. Participants will be stratified by age (18-59 years, ≥ 60 years) and study sites (if applicable).

For efficacy visits, study staff will contact participants on a weekly basis to remind reporting any signs or symptoms of COVID-19. If participants report any signs or symptoms that may be related to COVID-19, they will be required to immediately conduct an unscheduled visit under the instruction by site staff for COVID-19 related assessment and receiving treatment as deemed appropriate.

For reactogenicity and safety visits, all vaccinated participants will be observed for 30 minutes after each dose vaccination at study site for solicited or unsolicited AEs, and will be given subject diary to record solicited AEs within 7 days after each vaccination, and unsolicited AEs from the 1st vaccination to 28 days after the 3rd vaccination.

Approximately 600 participants will be included in the immunogenicity subgroup. Except for the efficacy and safety follow-up visits described above, this subgroup will be collected blood sample on Day 0 (pre-vaccination) and 14 days (+3 days), 90 days (±15 days) and 6 months (±15 days) after the 3rd dose.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and older.
2. Able and willing to comply with all study requirements.
3. Willing to allow investigators to discuss the medical history with his/her general practitioner/personal doctors and access all medical records which are relevant to study procedures.
4. Healthy adults, or adults with stable medical condition who have a pre-existing medical condition that does not meet any exclusion criteria. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
5. For females of childbearing potential only, willing to practice continuous effective contraception until 90 days after the final dose vaccination, and have negative pregnancy tests before each dose vaccination.

   * Nonchildbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or postmenopausal. A follicle-stimulating hormone (FSH) level and the amenorrhea duration (e.g. amenorrhea for ≥ 12 consecutive months prior to screening without an alternative medical cause) may be measured at the discretion of investigator to confirm postmenopausal status.
   * The effective contraceptive methods include sexual abstinence or adequate contraceptive measures such as intrauterine or implanted contraceptive device, oral contraceptives, injected or implanted contraceptives, sustained-release topical contraceptives, condoms (male), diaphragm, and cervical cap, etc.
6. Males participating in this study who are involved in heterosexual sexual activity must agree to practice adequate contraception (as described above) and refrain from donating sperm until 90 days after receiving the final dose vaccination.
7. Agreement to refrain from blood donation during the study.
8. Provide written informed consent form (ICF) prior to study enrollment.

Exclusion Criteria:

1. Laboratory confirmed SARS-CoV-2 infection defined by RT-PCR assay at screening. Participants with negative result for rapid antigen testing can be enrolled before having the result of RT-PCR assay, however, the participant needs to be withdrawn the following vaccination if the RT-PCR result shows positive.
2. SARS-CoV-2 antibodies (IgM or IgG) positive at screening.
3. Medical history of severe acute respiratory syndrome (SARS), middle east respiratory syndrome (MERS) and COVID-19 within 6 months prior to the randomization.
4. Fever (oral temperature ≥ 37.5°C / axillary temperature ≥ 37.3°C) on the day of vaccination or within recent 72 hours.
5. History of severe allergic disease or reactions likely to be exacerbated by any component of ReCOV, such as allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopaenic purpura, local hypersensitive necrosis reaction (Arthus reaction), or prior history of serious adverse reaction to any vaccine or drug, such as allergy, urticaria eczema, dyspnea, and angioneurotic edema.
6. Have malignant tumor (except for skin basal cell carcinoma or carcinoma uterine cervix in situ) and immune disease (e.g., documented human immunodeficiency virus [HIV] infection, systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy, and other immune disease that may influence immune response at investigator's discretion).
7. Have other severe and/or uncontrolled conditions, including but not limited to, acute infectious disease, cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, hematology disease, endocrine disorder, psychiatric condition and neurological illness. Uncontrolled condition is defined as significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
8. Have bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venipuncture.
9. Received immunosuppressant or other immunomodulators, antiallergic therapy, or cytotoxicity therapy for 14 or more consecutive days within 6 months before receiving the investigational product (IP). Local administration of immunosuppressant or immunomodulator is allowed (e.g., ointment, eye drops, inhalation, or nasal spray). Drugs for local administration should not be given at a dose over the recommended level in package insert or participants should have no signs of systemic exposure.
10. Administration of immunoglobulin and/or blood product within 3 months before using the IP or plan to use that during the study.
11. Continuous use of anticoagulants, such as coumarins and related anticoagulants (i.e., warfarin) or novel oral anticoagulants (i.e., apixaban, rivaroxaban, dabigatran and edoxaban).
12. Used other investigational drug or interventional device within 1 month before using the IP or plan to use that during the study, or are using other investigational drug or are within 5 half-lives after the last dose of the investigational drug.
13. Used subunit or inactivated vaccine within 14 days before using the IP, or used attenuated live or mRNA vaccine within 1 months (30 days) before using the IP, or plan to receive any other vaccines (except for the seasonal influenza vaccine, or emergency use authorized vaccines) during the study.
14. Prior receipt of an investigational or licensed COVID-19 vaccine, or investigational or approved vaccine against a coronavirus, including but not limited to SARS-CoV-1 and MERS-CoV.
15. Suspected or known current alcohol or drug dependency.
16. Pregnancy, lactation or willingness/intention to become pregnant within 90 days after receiving the last dose of study vaccine.
17. Staff of study site, the sponsor, and contract research organization (CRO) taking part in study conduct.
18. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data at investigator's discretion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7623 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of ReCOV in preventing Reverse Transcription-Polymerase Chain Reaction (RT-PCR) confirmed symptomatic COVID-19 in adults | > 14 days after 3 doses vaccination.
  RT-PCR confirmed symptomatic COVID-19 cases (regardless of severity) that occurred > 14 days after 3 doses vaccination.

SECONDARY OUTCOMES:
Evaluate the safety and reactogenicity | within 7 days after each vaccination
  The occurrence of solicited local and systemic adverse events (AEs) within 7 days after each vaccination.
Evaluate the safety and reactogenicity | from the 1st dose to 28 days after the 3rd vaccination.
  The occurrence of unsolicited AEs from the 1st dose to 28 days after the 3rd vaccination
Evaluate the safety and reactogenicity | from the 1st dose to the end of study.
  The occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs) from the 1st dose to the end of study.
To evaluate the efficacy of ReCOV in preventing RT-PCR confirmed symptomatic COVID-19 with various severity in adults | > 14 days after 3 doses vaccination.
  RT-PCR confirmed moderate, severe, critical COVID -19, or death that occurred > 14 days after 3 doses vaccination
To evaluate the efficacy of ReCOV in preventing RT-PCR confirmed symptomatic COVID-19 with various severity in adults | > 14 days after 3 doses vaccination.
  RT-PCR confirmed severe, critical COVID-19, or death that occurred > 14 days after 3 doses vaccination.
To evaluate the efficacy of ReCOV in preventing RT-PCR confirmed symptomatic COVID-19 with various severity in adults | > 14 days after 3 doses vaccination in different age groups (18-59 years and ≥ 60 years ).
  RT-PCR confirmed symptomatic COVID-19 cases (regardless of severity) that occurred > 14 days after 3 doses vaccination in different age groups (18-59 years and ≥ 60 years ).
To evaluate the immunogenicity of ReCOV | at 14 days, 3 months and 6 months after 3 doses vaccination
  The seroconversion rate (SCR), geometric mean titer (GMT) and geometric mean increase (GMI) of neutralizing antibody against prototype and epidemic strain at 14 days, 3 months and 6 months after 3 doses vaccination.
To compare the immunogenicity of ReCOV between Asian and Non-Asian in the immunogenicity subgroup | at 14 days,3 months and 6 months after 3 doses vaccination
  The SCR and GMT of neutralizing antibody against prototype at 14 days,3 months and 6 months after 3 doses vaccination.
Genotyping of SARS-CoV-2 virus nucleic acid sequence of COVID-19 cases to evaluate the possible viral mutations | >14 days after 3 doses vaccination
  SARS-CoV-2 virus nucleic acid sequence of RT-PCR confirmed symptomatic COVID-19 cases that occurred >14 days after 3 doses vaccination derived from isolates or direct nasopharyngeal (NP) (preferred)/ oropharyngeal (OP) swab, or respiratory samples (including saliva samples, or bronchoalveolar lavage fluid, if applicable).

OTHER OUTCOMES:
Exploratory : | > 14 days after the first dose vaccination
  To evaluate the efficacy of ReCOV after the first dose vaccination in preventing RT-PCR confirmed symptomatic COVID-19 in adults aged 18 years and older.

CONTACTS AND LOCATIONS:
Locations (11):
- B.P. Koirala Institute of Health Sciences, Dharān, Nepal
- Russia (10):
  - Aramil City Hospital, Aramil
  - LLC Medical Service solutions, Izhevsk
  - 'Federal State Budgetary Scientific Institution "Russian Scientific Centre of Surgery named after academician B.V. Petrovsky", Moscow
  - 'Joint Stock Company "Clinical and diagnostic center "Euromedservice", Moscow
  - State Regional Budgetary Institution of Healthcare "Murmansk Regional Clinical Hospital named after P.A. Bayandin", Murmansk
  - LLC Professorskaya klinika, Perm
  - UZI 4D Clinic LLC, Pyatigorsk
  - Klinika Zvyezdnaya LLC, Saint Petersburg
  - Limited Liability Company "Sfera-Med", Saint Petersburg
  - Research Center Eco-safety, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available